CLINICAL TRIAL: NCT01526980
Title: A Single-Centre, Randomised, Open-Labelled, Two-Period, Crossover Trial In Subjects With Type 2 Diabetes Comparing the Glycaemic Control of Two Treatment Regimens: A Thrice Daily Regimen With Biphasic Insulin Aspart 70 and - 30 and a Twice Daily Regimen With Biphasic Human Insulin 30
Brief Title: Glycaemic Control of Biphasic Insulin Aspart 70 and 30 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1319
Record Dates: First submitted 2012-02-01; First posted 2012-02-06 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; biphasic human insulin 30

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment period 1 (Experimental)
  Interventions: Drug: biphasic insulin aspart 30; Drug: biphasic insulin aspart 70; Drug: biphasic human insulin 30
- Treatment period 2 (Active Comparator)
  Interventions: Drug: biphasic insulin aspart 30; Drug: biphasic insulin aspart 70; Drug: biphasic human insulin 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Administrated subcutaneously (s.c., under the skin) once daily before dinner for 30 days in each treatment period
Drug: biphasic insulin aspart 70 — Administrated subcutaneously (s.c., under the skin) twice daily before breakfast and lunch for 30 days in each treatment period
Drug: biphasic human insulin 30 — Administrated subcutaneously (s.c., under the skin) twice daily before breakfast and dinner for 30 days in each treatment period

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare the glycaemic control of biphasic insulin aspart 70 + biphasic insulin aspart 30 with biphasic human insulin 30 in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type 2 diabetes
* Treatment with BHI (biphasic human insulin) 30 twice daily for at least three months
* HbA1c maximum 10.0%
* BMI (Body Mass Index) maximum 35.0 kg/m2
* Able and willing to perform self-blood glucose monitoring (SBGM)

Exclusion Criteria:

* The receipt of any investigational drug within the last 30 days prior to this trial
* Total daily insulin dose minimum 2.0 U/(kg·day)
* A history of drug abuse or alcohol dependence within the last 5 years
* Impaired hepatic function
* Impaired renal function
* Cardiac disease
* Severe, uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2002-05; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Glucose average in 24-hour blood glucose profiles

SECONDARY OUTCOMES:
Pre-meal glucose level
Post-meal excursion of glucose (0-4 hours)
Cmax, maximum concentration of total insulin
tmax, time of maximum concentration of total insulin
The area under the 24-hour total insulin concentration time curve
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Newcastle, United Kingdom

REFERENCES:
- [Result] Dashora U, Ashwell SG, Home PD. An exploratory study of the effect of using high-mix biphasic insulin aspart in people with type 2 diabetes. Diabetes Obes Metab. 2009 Jul;11(7):680-7. doi: 10.1111/j.1463-1326.2008.01024.x. PMID 19527481
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com